CLINICAL TRIAL: NCT01598597
Title: An Observational Pilot Study Evaluating the Feasibility of Conducting Genome-Wide Association Studies Utilizing Subject Provided Information in Subjects With Locally Recurrent or Metastatic Breast Cancer, Metastatic Colorectal Cancer, Metastatic Non-Squamous Non-Small Cell Lung Cancer, Recurrent Glioblastoma, or Metastatic Renal Cell Cancer Treated With Avastin
Brief Title: An Observational Pilot Study Evaluating the Feasibility of Conducting Genome-Wide Association Studies Utilizing Subject Provided Information in Subjects With Locally Recurrent or MBC, MCRC, MNSCLC, RGBM or MRCC Treated With Avastin (Bevacizumab) (InVite)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Collaborators: 23andMe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GO28289
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Colorectal Cancer; Non-Small Cell Lung Cancer; Glioblastoma; Renal Cell Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Glioblastoma; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, optional blood

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This pilot, non-interventional, observational, Web-based, prospective cohort study is designed to collect self-reported safety and effectiveness and genetic data from subjects with locally recurrent breast cancer (BC) or metastatic breast cancer (MBC), metastatic colorectal cancer (MCRC), metastatic non-squamous non-small cell lung cancer (MNSCLC), recurrent glioblastoma (RGBM), or metastatic renal cell cancer (MRCC) in the United States who have been previously treated with Avastin (bevacizumab). The cohort will be composed of male and female subjects who have been diagnosed with locally recurrent BC or MBC, MCRC, MNSCLC, RGBM, or MRCC who have received treatment with bevacizumab in combination with chemotherapy, which started prior to or up to 31 December 2012. Participants will be self-referred to this study. They will be recruited online via a number of sources, including through the involvement of patient advocacy groups, social media tools, traditional media, physicians, and events to raise awareness of this study. After appropriate informed consent and authorization are obtained, data will be collected directly from subjects in an online survey. Participants will be contacted electronically to complete quarterly follow-up surveys. The follow-up period will be 1 year from responding to the baseline survey. DNA collection will be performed as part of this study. DNA will be extracted from saliva, which will be provided by the subject utilizing a collection kit sent to the participants for at-home use.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent BC or MBC, MCRC, MNSCLC, RGBM, or MRCC in patients treated or on treatment with bevacizumab, which started prior to or up to 31 December 2012
* Ability to read and understand English
* Ability to access and use a computer connected to the Internet
* Signed informed consent and authorization form
* Residence in the United States
* At least 18 years of age

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with history of metastatic or locally recurrent breast cancer treated with Avastin
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who complete the survey and who provide evaluable genetic information (DNA) | 24 months

SECONDARY OUTCOMES:
Clinical characteristics (current disease status/previous treatments) of subjects participating in this study | 24 months
Demographic distribution (age, sex) of subjects participating in this study | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (50):
- United States (50):
  - Many Locations, Alabama
  - Many Locations, Alaska
  - Many Locations, Arizona
  - Many Locations, Arkansas
  - Many Locations, California
  - Many Locations, Colorado
  - Many Locations, Connecticut
  - Many Locations, Delaware
  - Many Locations, Florida
  - Many Locations, Georgia
  - Many Locations, Hawaii
  - Many Locations, Idaho
  - Many Locations, Illinois
  - Many Locations, Indiana
  - Many Locations, Iowa
  - Many Locations, Kansas
  - Many Locations, Kentucky
  - Many Locations, Louisiana
  - Many Locations, Maine
  - Many Locations, Maryland
  - Many Locations, Massachusetts
  - Many Locations, Michigan
  - Many Locations, Minnesota
  - Many Locations, Mississippi
  - Many Locations, Missouri
  - Many Locations, Montana
  - Many Locations, Nebraska
  - Many Locations, Nevada
  - Many Locations, New Hampshire
  - Many Locations, New Jersey
  - Many Locations, New Mexico
  - Many Locations, New York
  - Many Locations, North Carolina
  - Many Locations, North Dakota
  - Many Locations, Ohio
  - Many Locations, Oklahoma
  - Many Locations, Oregon
  - Many Locations, Pennsylvania
  - Many Locations, Rhode Island
  - Many Locations, South Carolina
  - Many Locations, South Dakota
  - Many Locations, Tennessee
  - Many Locations, Texas
  - Many Locations, Utah
  - Many Locations, Vermont
  - Many Locations, Virginia
  - Many Locations, Washington
  - Many Locations, West Virginia
  - Many Locations, Wisconsin
  - Many Locations, Wyoming